CLINICAL TRIAL: NCT03546205
Title: A Single-dose, Open-label, Parallel-group Study to Evaluate JNJ-64565111 Pharmacokinetics and Safety in Adult Subjects With Varying Degrees of Renal Function
Brief Title: A Study to Evaluate JNJ-64565111 Pharmacokinetics and Safety in Adult Participants With Varying Degrees of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108474; 64565111OBE1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: JNJ-64565111 (Experimental): Participants with normal renal function and no evidence of kidney damage (estimated glomerular filtration rate [eGFR] greater than or equal to [>=] 90 milliliter/minute [mL/min]) will be enrolled. Participants will receive a single subcutaneous (SC) dose of JNJ-64565111 on Day 1.
  Interventions: Drug: JNJ-64565111
- Group 2: JNJ-64565111 (Experimental): Participants with mild renal impairment (eGFR 60 to less than [<] 90 mL/min) will be enrolled. Participants will receive a single SC dose of JNJ-64565111 on Day 1.
  Interventions: Drug: JNJ-64565111
- Group 3: JNJ-64565111 (Experimental): Participants with moderate renal impairment (eGFR 30 to <60 mL/min) will be enrolled. Participants will receive a single SC dose of JNJ-64565111 on Day 1.
  Interventions: Drug: JNJ-64565111
- Group 4: JNJ-64565111 (Experimental): Participants with severe renal impairment (eGFR <30 mL/min) will be enrolled. Participants will receive a single SC dose of JNJ-64565111 on Day 1.
  Interventions: Drug: JNJ-64565111
- Group 5: JNJ-64565111 (Experimental): Participants with end-stage renal disease (requiring hemodialysis 3 times per week for at least 3 months before screening; eGFR will not be calculated) will be enrolled. Participants will receive a single SC dose of JNJ-64565111 on Day 1.
  Interventions: Drug: JNJ-64565111

INTERVENTIONS:
Drug: JNJ-64565111 — All participants will receive a single SC dose of JNJ-64565111 solution on Day 1.

SUMMARY:
The purpose of study is to evaluate the pharmacokinetics of a single, subcutaneous dose of JNJ-64565111 in adult participants with varying degrees of renal function including participants with end stage renal disease, requiring hemodialysis, compared with participants with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* If a woman, must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, or if sexually active, be practicing an effective method of birth control before entry and throughout the study
* A woman must have a negative highly sensitive serum (beta human chorionic gonadotropin [hCG]) at screening. On Day -1, female non-end-stage renal disease (ESRD) participants should have a negative urine pregnancy test and female ESRD participants requiring hemodialysis (HD) should have a negative serum pregnancy test
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction (from screening through Day 42 postdose)
* Body mass index (weight [kilogram {kg}]/height^2 [ meter {m}]^2) between 18 and 40 kg/m^2 (inclusive), and body weight not less than 50 kg
* Have normal renal function defined as: predicted estimated glomerular filtration rate greater than or equal to (>=) 90 milliliter (mL)/minute based on the Chronic Kidney Disease-Epidemiology formula (for participants with normal renal function)

Exclusion Criteria:

* History of, or a reason to believe a participant has a history of, drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM V) criteria within 5 years before screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, opiates, opioids, cocaine, cannabinoids, amphetamines, and benzodiazepines) at screening and Day -1 of the treatment period (unless medically prescribed)
* Any surgical or medical condition that potentially may alter the absorption, metabolism, or excretion of the study drug, with the exception of renal impairment as described in the inclusion criteria, and except for participants who had a cholecystectomy or a hernia repair
* History of clinically significant allergies, especially known hypersensitivity or intolerances
* Known allergy to JNJ-64565111 or its excipients
* Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study or at least 2 months after the completion of the study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Analyte Concentration (Cmax) of JNJ-64565111 | Predose, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 984 hours postdose
  Cmax is the maximum observed serum analyte concentration of JNJ-64565111.
Area Under the Serum Analyte Concentration-Time Curve from Time Zero to Last Measurable (not Below Quantification Limit) Concentration (AUC[0-last]) of JNJ-64565111 | Predose, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 984 hours postdose
  AUC [0-Last] is the area under the serum analyte concentration versus time curve from time zero to the time of the last measurable (not below quantification limit) concentration of JNJ-64565111, calculated by linear-linear trapezoidal summation.
Area Under the Serum Analyte Concentration-Time Curve from Time Zero to Infinite Time (AUC[0-infinity]) of JNJ-64565111 | Predose, 4, 8, 12, 24, 36, 48, 72, 96, 144, 216, 384, 672, and 984 hours postdose
  AUC (0-infinity) is the area under the serum analyte concentration-time curve from time zero to infinite time, calculated as AUC(last) + C(last)/lamda(z) where C(last) is the last observed measurable (not below quantification limit) concentration of JNJ-64565111.

SECONDARY OUTCOMES:
Number of Participants with Antibodies to JNJ-64565111 | Predose, Days 7, 29 and 42
  Number of participants with antibodies to JNJ-64565111 will be reported.
Number of Participants with Adverse Events | Approximately 9 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily have a causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - AMR New Orleans, Formerly New Orleans Center for Clinical Research - New Orleans, an AMR company, Knoxville, Tennessee